CLINICAL TRIAL: NCT06675669
Title: The Effect of Reflective Thinking Method Used in Ethics Teaching on Ethical Decision Making, Professional Values and Compassion Level in Nursing Students
Brief Title: Effect of Reflective Thinking Method on Ethical Decision Making, Professional Values and Compassion Level
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Serpil SU, Principal Investigator, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: NecErbakanU
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Ethical Decision Making; Professional Values; Compassion
Keywords: reflective thinking; ethics teaching; ethical decision making; professional values; compassion; nursing students

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reflective thinking (Experimental): Discussion sessions will be held once a week for 7 weeks within the scope of the Professional Ethics Course for the students in the intervention group. For the discussion sessions, the students will be divided into 4 groups of 10-11 people. Separate 1-hour discussion sessions will be held with each group.
  A training session will be held with the students in the intervention group in the first week (November 22,2024). In this session; the researchers will inform the students about the reflective thinking technique. In the 2nd, 3rd, 4th, 5th, 6th and 7th weeks (January 03, 2025), the students will come to class by writing an event/situation they encountered during their hospital internship in the Obstetrics and Gynecology Nursing course, which they are currently doing clinical practice. During the class hour, the researcher will determine one of the events/situations written by the students and will discuss it in the group.Follow-up data will be collected after 3 months (March 31,2025).
  Interventions: Other: Reflective thinking method
- Control (No Intervention): No application will be made to the students in the control group. These students will be given standard education for 7 weeks (Between November 22, 2024 and January 03, 2025).

INTERVENTIONS:
Other: Reflective thinking method — It will be applied to students in the initiative group for 1 hour per week for 7 weeks.
  Arms: Reflective thinking

SUMMARY:
This randomized controlled study aimed to determine the effect of the reflective thinking method used in ethics education on ethical decision making, professional values, and compassion levels in nursing students.The hypotheses of the study are as follows:

H1.1. There is a difference in ethical decision-making average scores between students who were applied the reflection method in ethics education and students in the control group.

H1.2. There is a difference in professional values average scores between students who were applied the reflection method in ethics education and students in the control group.

H1.3. There is a difference in compassion average scores between students who were applied the reflection method in ethics education and students in the control group.

DETAILED DESCRIPTION:
The research will be conducted as a pre-test-post-test, parallel group randomized controlled experimental design. The sample of the research to be conducted at Necmettin Erbakan University Faculty of Nursing consists of 84 students. Students who meet the inclusion criteria will be assigned to the intervention and control groups by the block randomization method. The intervention group will be given ethics training with the reflective thinking method, while the control group will be given standard ethics training. The research data will be collected between November 22, 2024 and March 31, 2025 using the Student Information Form, Nursing Ethical Dilemma Test, Professional Values Scale and Compassion Scale.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Being registered in the Professional Ethics course
* Having participated in the theoretical part of the Professional Ethics course
* Being volunteering to participate in the research

Exclusion Criteria:

* Having taken the Professional Ethics course before
* Working as a healthcare professional
* Being a foreign national

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-11-22 (Estimated); Primary Completion 2024-11-22 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Ethical Dilemma Test to determine the level of ethical decision making | 1st measurement will be made at week 1 (November 22, 2024); 2nd measurement at week 7 (January 03, 2025), 3rd follow-up measurement at week 19 (3 months later, March 31, 2025 ).
  The aim of determining the levels of "Principle Thinking" (F) and "Practical Thinking (P) is to determine the situation of encountering an ethical dilemma (Familiarity). The lowest "Principle Thinking" score that can be achieved in the test is 18, the highest "Principle Thinking" score is 66. The lowest "Practical Thinking" score that can be achieved is 6, and the highest "Practical Thinking" score is 36. In the familiarity section, 6-17 points indicate familiarity with a similar dilemma, and 18-30 points indicate unfamiliarity. High scores indicate a high level of ethical decision-making skills.

SECONDARY OUTCOMES:
Professional Values Scale for Nurses to determine the level of professional values | 1st measurement will be made at week 1 (November 22, 2024); 2nd measurement at week 7 (January 03, 2025), 3rd follow-up measurement at week 19 (3 months later, March 31, 2025 ).
  The lowest score that can be obtained from the scale is 26 and the highest score that can be obtained is 130. High scores indicate high professional values.
Compassion Scale to determine the level of compassion | 1st measurement will be made at week 1 (November 22, 2024); 2nd measurement at week 7 (January 03, 2025), 3rd follow-up measurement at week 19 (3 months later, March 31, 2025 ).
  The minimum score on the scale is 1 and the maximum score is 5. As the total score on the scale increases, the level of compassion also increases.

IPD SHARING:
Plan to Share IPD: No